CLINICAL TRIAL: NCT05857072
Title: Evaluation of the Mechanisms of Weight-bearing of the Hemiplegic Limb During Table Tennis Sessions in the Framework of Post-stroke Rehabilitation : Pilot Study
Acronym: HEMITENNIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: FondationbHopale (Other)
Responsible Party: Sponsor
Other Study IDs: HOP22-RIPH3-08
Record Dates: First submitted 2023-04-27; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Post-stroke; Hemiplegic Gait; Rehabilitation
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an experimental, observational, prospective study designed to develop medical knowledge.

The primary objective of the study is to analyze the weight bearing of the hemiplegic side according to the different areas of interest during the practice of table tennis.

This study is part of a usual framework of management of post-stroke hemiplegic patients with an additional passage to the movement laboratory to collect additional data collection, via the use of force plateforms, considered here as non-interventional.

The passage to the movement laboratory consists in the practice of a table tennis session including three game situations. Before to the table tennis session, the subject placed on the force plateforms, performs a spontaneous bipodal station followed by a maximum voluntary support transfer on the hemiplegic limb. During the table tennis session, the subject is filmed and his load on the hemiplegic side during the game situations is evaluated using the force platforms.

In addition of the table tennis session three questionnaires are administered to the patient in order to know :

* The static and dynamic balance in order to identify persons at risk of falling: Berg Balance and Evaluation Scale
* The degree of autonomy of the patient: Modified Rankin Score
* The Stroke severity: NIHSS score

ELIGIBILITY:
Inclusion Criteria:

* Patients treated at the Hopale Foundation for a stroke rehabilitation program
* Patients following the balance and coordination protocol - Minimum age of 18 years
* BERG score >40
* Subject has played table tennis at least once prior to the stroke.
* Patient is a member or beneficiary of a social security plan.
* Patient who has received informed information about the study and has given his/her consent
* Ability to understand French instructions.

Exclusion Criteria:

* Cognitive disorders notified in the medical file
* Subject under judicial protection :

  * Subject under guardianship
  * Subject under curatorship
  * Subject under protective measure
* Pregnant or breastfeeding woman
* Patient with cognitive disorders preventing the comprehension of instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited among the patients included in the "balance and coordination" rehabilitation protocol at the Jacques Calvé center of the Hopale Foundation.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
To analyze the weight bearing on the hemiplegic side according to the different areas of interest of interest during the practice of table tennis. | During the only table tennis session on the one day of patient inclusion
  The vertical force peaks (Fz) under the hemiplegic foot and under the non-injured foot recorded during the subject's ball returns throughout the session. These peaks will be categorized according to the zones and the shots used by the subject.

SECONDARY OUTCOMES:
To compare the weight bearing on the hemiplegic side during table tennis practice to a voluntary weight-bearing exercise on the injured limb. | During the only table tennis session on the one day of patient inclusion
  Peak vertical force (Fz) under the hemiplegic foot and under the non-injured foot are compared between table tennis and the analytical exercise of voluntary weight-bearing voluntary.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie PERSINE, Principal Investigator — Centre Calvé, Fondation Hopale
Locations (1):
- Institut Calvé, Berck, France

REFERENCES:
- See also: Related Info — https://doi.org/10.1016/j.annrmp.2004.04.004
- See also: Related Info — https://europepmc.org/article/med/34824919
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30362890/
- See also: Related Info — https://www.em-consulte.com/article/749535/troubles-statiques-de-lhemiplegique-evaluation-sur